CLINICAL TRIAL: NCT00865020
Title: A Twelve-week, Randomized, Double-blind, Parallel Group Study to Evaluate the Prolonged Efficacy and Safety of Aliskiren 300 mg Compared to Telmisartan 80 mg in Mild to Moderate Hypertensive Patients With the 24-hour Ambulatory Blood Pressure Measurement After 1 Week of Treatment Withdrawal Study Acronym: ASSERTIVE - AliSkiren Study of Profound antihypERtensive Efficacy in hyperTensIVE Patients
Brief Title: Efficacy and Safety of Aliskiren 300 mg Compared to Telmisartan 80 mg After 1 Week of Treatment Withdrawal
Acronym: ASSERTIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2408
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: Hypertension; ABPM; systolic blood pressure; diastolic blood pressure; cardiovascular disease; aliskiren; telmisartan
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — aliskiren; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aliskiren 300 mg (Experimental): Aliskiren tablets starting at a dose of 150 mg taken orally daily for 2 weeks followed by a dose of 300 mg taken orally for 10 weeks and placebo (withdrawal) for one week. Participants took Placebo to Aliskiren: 1 tablet for the first 2 weeks and 2 tablets during the one week withdrawal period.
  Interventions: Drug: Aliskiren; Drug: Placebo to Aliskiren
- Telmisartan 80 mg (Active Comparator): Telmisartan capsules starting at a dose of 40 mg taken orally daily for 2 weeks followed by a dose of 80 mg taken orally daily for 10 weeks and placebo (withdrawal) for one week. Participants took Placebo to Telmisartan: 1 capsule for the first 2 weeks and 2 capsules during the one week withdrawal period.
  Interventions: Drug: Telmisartan; Drug: Placebo to Telmisartan

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg tablets taken orally daily. 1 tablet for the first two weeks followed by 2 tablets for 10 weeks.
  Arms: Aliskiren 300 mg
Drug: Telmisartan — Telmisartan 40 mg capsules taken orally daily. 1 capsule the first 2 weeks followed by 2 capsules for 10 weeks.
  Arms: Telmisartan 80 mg
Drug: Placebo to Aliskiren — Placebo to Aliskiren tablets taken orally daily. 1 Tablet for the first 2 weeks and 2 tablets during the no treatment (withdrawal) week.
  Arms: Aliskiren 300 mg
Drug: Placebo to Telmisartan — Placebo to Telmisartan capsule taken orally daily. 1 capsule for the first 2 weeks and 2 capsules during the no treatment (withdrawal) week.
  Arms: Telmisartan 80 mg

SUMMARY:
This study was specifically designed to provide additional information on the mechanism of action of direct renin inhibition postulating the higher-level RAS cascade inhibition. The purpose of this study was to compare the prolonged efficacy and safety of aliskiren to that of telmisartan in mild to moderate hypertensive patients in the 24 hrs Ambulatory Blood Pressure Monitoring setting after a one week treatment withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Mean sitting systolic blood pressure ≥ 140 mmHg and < 180 mmHg
* 24-hr mean ambulatory systolic blood pressure ≥ 135 mmHg

Exclusion Criteria:

* Severe hypertension defined as mean sitting systolic blood pressure ≥ 180 mmHg and/or mean sitting diastolic blood pressure ≥ 110 mmHg
* Patients with Type 1 diabetes mellitus
* Secondary hypertension of any etiology
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (16):
- Investigative Site, Sorocaba, Brazil
- Investigative Site, Gatineau, Canada
- Investigative Site, Guayaquil, Ecuador
- Investigative Site, Erfurt, Germany
- Invesitagtive Site, Budapest, Hungary
- Investigative Site, Kuala Lumpur, Malaysia
- Investigative Site, Mexico City, Mexico
- Investigative Site, Panama City, Panama
- Investigative Site, Manila, Philippines
- Investigative Site, Singapore, Singapore
- Investigative Site, Bratislava, Slovakia
- Investigative Site, Cheongju-si, South Korea
- Investigative Site, Seville, Spain
- Investigative Site, Istanbul, Turkey (Türkiye)
- Investigative Site, Westbury, United Kingdom
- Investigative Site, Caracas, Venezuela

REFERENCES:
- [Derived] Wang GM, Li LJ, Fan L, Xu M, Tang WL, Wright JM. Renin inhibitors versus angiotensin receptor blockers for primary hypertension. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD012570. doi: 10.1002/14651858.CD012570.pub2. PMID 40013543
- [Derived] Williams B, Lacy PS, Baschiera F, Brunel P, Dusing R. Novel description of the 24-hour circadian rhythms of brachial versus central aortic blood pressure and the impact of blood pressure treatment in a randomized controlled clinical trial: The Ambulatory Central Aortic Pressure (AmCAP) Study. Hypertension. 2013 Jun;61(6):1168-76. doi: 10.1161/HYPERTENSIONAHA.111.00763. Epub 2013 Apr 29. PMID 23630950
- [Derived] Dusing R, Brunel P, Baek I, Baschiera F. Sustained blood pressure-lowering effect of aliskiren compared with telmisartan after a single missed dose. J Clin Hypertens (Greenwich). 2013 Jan;15(1):41-7. doi: 10.1111/jch.12018. Epub 2012 Oct 9. PMID 23282123

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1359 participants entered the Placebo Run-In phase which was 1-2 weeks in duration. Those participants completing the Placebo-Run-In Phase were randomized to receive either aliskiren 300 mg or telmisartan 80 mg.
Period: Overall Study
Arm/Group | Aliskiren 300 mg | Telmisartan 80 mg
Started | 414 | 408
Completed | 365 | 357
Not Completed | 49 | 51
Not completed — Withdrawal by Subject | 22 | 16
Not completed — Adverse Event | 9 | 14
Not completed — Abnormal test procedure result(s) | 6 | 8
Not completed — Lost to Follow-up | 6 | 4
Not completed — Protocol deviation | 4 | 1
Not completed — Administrative problems | 0 | 2
Not completed — Abnormal laboratory value(s) | 0 | 1
Not completed — Death | 0 | 1
Not completed — Randomized but discontinued | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren 300 mg | Telmisartan 80 mg | Total
Number analyzed (Participants) | 414 | 408 | 822
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.46) | 56.0 (11.91) | 55.9 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 178 | 384
  Male | 208 | 230 | 438

OUTCOME MEASURES:

1. Primary Outcome: Change in 24 Hour (24-Hr) Mean Ambulatory Systolic Blood Pressure (MASBP) From the End of the Active Treatment Period to Day 7 of the Withdrawal Period
Description: An Ambulatory Blood Pressure Monitor measured a participants's blood pressure over a 24 hour period using an automated validated monitoring device at week 12 (end of the active treatment) and at week 13 (end of the day 7 withdrawal period). The 24 Hour MASBP was calculated by taking the mean of all Ambulatory Systolic Blood Pressure readings for the 24 hour period. The difference of the 24 hour MASBP from the end of the active treatment to Day 7 of the treatment withdrawal period was calculated using a two way analysis of variance with treatment and region as factors.
Time Frame: 12 weeks, 13 weeks
Population: ABPM Completer Set consisting of all participants in the Full Analysis set who had ABPM measurements at the end of the active treatment period and Day 7 of the treatment withdrawal period.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren 300 mg | Telmisartan 80 mg
Number analyzed (Participants) | 330 | 336
mmHg | 2.70 (0.466) | 6.51 (0.461)

2. Secondary Outcome: Change in 24 Hour (24-hr) Mean Ambulatory Diastolic Blood Pressure (MADBP) From the End of the Active Treatment Period to Day 7 of the Withdrawal Period
Description: An Ambulatory Blood Pressure Monitor measured a participants's blood pressure over a 24 hour period using an automated validated monitoring device at week 12 (end of the active treatment) and at week 13 (end of the day 7 withdrawal period). The 24 Hour MADBP was calculated by taking the mean of all Ambulatory Diastolic Blood Pressure readings for the 24 hour period. The difference of the 24 hour MADBP from the end of the active treatment to Day 7 of the withdrawal period was calculated using a two way analysis of variance with treatment and region as factors.
Time Frame: 12 weeks, 13 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren 300 mg | Telmisartan 80 mg
Number analyzed (Participants) | 330 | 336
mmHg | 2.09 (0.328) | 4.21 (0.324)

3. Secondary Outcome: Change in 24-hr Mean Ambulatory Systolic Blood Pressure (MASBP) and Mean Ambulatory Diastolic Blood Pressure (MADBP) From Baseline to Day 7 of the Withdrawal Period
Description: An Ambulatory Blood Pressure Monitor measured a participants's blood pressure over a 24 hour period using an automated validated monitoring device at Baseline (at Randomization) and at week 13 (day 7 of the withdrawal period). The 4 Hour MASBP and MADBP was calculated by taking the mean of all Ambulatory Blood Pressure readings during the 24 hour period. The difference of the 24 hour measurements from baseline to day 7 of the withdrawal period were calculated using a two way analysis of variance with treatment and region as factors and baseline as a covariate.
Time Frame: Baseline, 13 weeks
Population: Full Analysis Set consisting of all participants randomized to treatment with measurements at baseline and day 7 of the withdrawal period.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren 300 mg | Telmisartan 80 mg
Number analyzed (Participants) | 336 | 339
mmHg
  MASBP | -8.39 (0.542) | -5.59 (0.539)
  MADBP | -5.05 (0.379) | -3.44 (0.377)

4. Secondary Outcome: Change in the Mean Sitting Systolic Blood Pressure (msSBP) as Measured at All Study Visits During the Double-blind Treatment Period and During the Treatment Withdrawal Period
Description: Blood Pressure was measured in the office after the patient was sitting for 5 minutes. The average of 3 readings 1-2 minutes apart were used in the analysis.
  The change in the double-blind period was calculated from the end of active treatment at week 12 to the Baseline (Randomization) using Analysis of Covariance with treatment and region as factors and baseline msSBP as a covariate.
  The change in the treatment interruption period was calculated from day 7 of the withdrawal period at week 13 to the end of the active treatment using Analysis of Variance with treatment and region as factors.
Time Frame: Baseline, 12 weeks, 13 weeks
Population: Full Analysis set consisting of all participants randomized to treatment. n1=participants with measurements at baseline and end of the active treatment period for the Double-blind Period. n2=participants with measurements at the end of the active treatment period and end of the treatment withdrawal period for the Treatment Interruption Period.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren 300 mg | Telmisartan 80 mg
Number analyzed (Participants) | 412 | 406
mmHg
  Double-Blind Period (n1=374,371) | -15.22 (0.744) | -14.64 (0.744)
  Treatment Interruption Period (n2=369,363) | 1.26 (0.652) | 5.00 (0.658)

5. Secondary Outcome: Change in the Mean Diastolic Sitting Blood Pressure (msDBP) as Measured at All Study Visits During the Double-blind Treatment Period and During the Treatment Withdrawal Period
Description: Blood Pressure was measured in the office after the patient was sitting for 5 minutes. The average of 3 readings 1-2 min. apart were used in the analysis.
  The change in the double-blind period was calculated from the end of active treatment at week 12 to the Baseline (Randomization) using Analysis of Covariance with treatment and region as factors and baseline msDBP as a covariate.
  The change in the treatment interruption period was calculated from day 7 of the withdrawal period at week 13 to the end of the active treatment using Analysis of Variance with treatment and region as factors.
Time Frame: Baseline, 12 weeks, 13 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren 300 mg | Telmisartan 80 mg
Number analyzed (Participants) | 412 | 406
mmHg
  Double-Blind Period (n1=374,371) | -6.35 (0.453) | -6.60 (0.453)
  Treatment Interruption Period (n2=369,363) | 0.03 (0.388) | 2.69 (0.392)

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: Safety Set consisting of all participants who received at least one dose of double-blind study treatment.
Arm/Group | Aliskiren 300 mg | Telmisartan 80 mg
Serious Adverse Events (participants affected / at risk) | 3/411 | 5/403
Other Adverse Events (participants affected / at risk) | 15/411 | 32/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (N=411) | Telmisartan 80 mg (N=403)
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (N=411) | Telmisartan 80 mg (N=403)
Headache (Nervous system disorders) | 15 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.